CLINICAL TRIAL: NCT00894491
Title: Complementary and Alternative Medical Therapy Trends: A Patient Survey in a University Based Clinic
Brief Title: Complementary and Alternative Medical Trends: A Patient Survey in a University Based Clinic
Status: Withdrawn | Type: Observational
Why Stopped: Nonapplicable clinical trial
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-4872
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Complementary and Alternative Therapies
Keywords: alternative medicine; complementary medicine; acupuncture; Chinese herbals

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Patient survey identifying key elements of patient experience and decision-making processes regarding attendance University of California, Irvine (UCI)'s Integrative Medicine Clinic.

DETAILED DESCRIPTION:
Patient survey to determine why patients come to UCI's integrative medicine clinic, whether they would prefer we accept insurance coverage, and what therapies they are using.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 41 years of age or older
* English speaking
* Ability to provide informed consent
* Patient at Gottschalk Medical Plaza Integrative Medical Clinic
* Ability to complete survey

Exclusion Criteria:

* Patient less than 41 years of age
* Inability to speak English
* Patient unable to provide informed consent
* Patient not being seen at Gottschalk medical Plaza Integrative Medical Clinic
* Incomplete survey

Min Age: 41 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 14 male, 19 female white non-Hispanic, college educated over the age of 41
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-05 (Actual); Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Why People Chose Complementary and Alternative Therapies | Post-care

CONTACTS AND LOCATIONS:
Overall Officials: John Longhurst, M.D., Ph.D., Principal Investigator — UC Irvine School of Medicine
Locations (1):
- UCI Samueli Center Clinic, Newport Beach, California, United States